CLINICAL TRIAL: NCT02412839
Title: Population Research of Sublingual Microcirculation Data of Healthy Volunteers by Using the Third Generation Microcirculation Video Microscope
Brief Title: Sublingual Microcirculation of Healthy Volunteers by Using the Third Generation Microcirculation Video Microscope
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201502027RIND
Record Dates: First submitted 2015-04-06; First posted 2015-04-09 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 20-39: Patients aged from 20 to 39 years old. 30 males and 30 females.
- Group 40-59: Patients aged from 40 to 59 years old. 30 males and 30 females.
- Group 60-79: Patients aged from 60 to 79 years old. 15 males and 15 females.

SUMMARY:
This study will enroll 150 healthy volunteers, and the grouping is as follows: group 20-39 (30 males and 30 females); group 40-59 (30 males and 30 females); and group 60-79 (15 males and 15 females). The sublingual microcirculation will be examined with the incident dark field video microscope (Cytocam，Braedius Battery Powered Transilluminator). The study aims to compare the differences of microcirculation among the three groups and between genders.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged from 20 to 79 years old
* BMI ranged from 18.5 to 27 kg/m2

Exclusion Criteria:

* Systolic blood pressure > 140 mm Hg, diastolic blood pressure > 95 mm Hg, or systolic blood pressure < 90 mm Hg at enrollment
* Body temperature > 37.5 ℃ or < 35.5 ℃ at enrollment
* had been diagnose with any one of the following diseases

  * hypertension
  * diabetes mellitus
  * peripheral arterial occlusive disease
  * coronary arterial disease
  * liver cirrhosis
  * chronic kidney disease
  * stroke
  * anemia
  * asthma
  * chronic bronchitis
  * any metabolic diseases
  * any hematologic disease
  * uncured cancer
  * chronic uncontrolled infection
  * other disease may limit daily activities
  * non-native speakers

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-04; Primary Completion 2017-02-15 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Total small vessel density of sublingual small vessels measured by Cytocam | Once at enrollment
  Total small vessel density will be measured by Cytocam

SECONDARY OUTCOMES:
Perfused small vessel density of sublingual small vessels measured by Cytocam | Once at enrollment
  Perfused small vessel density will be measured by Cytocam

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chang Yeh, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan